CLINICAL TRIAL: NCT05973760
Title: Dietary Assessment and Prevention of Hypertension in Nigeria
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leeds (Other)
Collaborators: Rivers State University Teaching Hospital (Unknown); Tertiary Education Trust Fund (TETFund) (Unknown)
Responsible Party: Principal Investigator, Michael A Zulyniak, Dr., University of Leeds
Other Study IDs: FREC 2023-0484-572; RSUTH/REC/2023316 (Other: Rivers State University Teaching Hospital, Nigeria)
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Hypertension; Blood Pressure
Keywords: diet; West Africa; nutrition; LMIC
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypertensive: Men or women previously diagnosed with hypertension
- Non-hypertensive: Men or women not previously diagnosed with hypertension

SUMMARY:
Contrary to North America and Europe, the prevalence of hypertension is rising in West Africa and, currently, there are no simple dietary assessment tools for clinicians to offer personalized dietary support to their patients. This study aims to:

1. Evaluate the feasibility and validate the a short dietary screening tool for hypertension for use in Nigerian clinics; and
2. Test the accuracy and estimate the potential value of the validated short dietary assessment tool in Nigeria clinics.

DETAILED DESCRIPTION:
Contrary to North America and Europe, the prevalence of hypertension is rising in West Africa. With a transition from whole foods to processed foods in Nigeria, diet is considered a key driver of hypertension. To combat this, the national nutritional guidelines in Nigeria were implemented but their translation into actionable tools for clinicians remains a challenge. Currently, there are no simple dietary assessment tools that are concise and suitable to be incorporated into clinical care without requiring extensive data analysis while still providing personalized dietary support to their patients. This study aims to deliver a clinically tested and validated short dietary assessment tool for clinicians, patients, and researchers across Nigeria to provide personalised dietary advice for patients with hypertension.

The study will be conducted in two phases: Phase 1 (n=75), will investigate the feasibility of the short FFQ and its agreement with 24-hour dietary recalls (3x) in a clinical setting in Nigeria. During the analysis of Phase 1 data, a scoring system will be developed based on the associations between individual food items in the FFQ and measures of hypertension. Phase 2 (n=50) will assess the acceptability of the FFQ and validate the association between the FFQ score and hypertension.

We anticipate that the development of a clinically tested and validated short food frequency questionnaire that will be ready for implementation analysis for use by clinicians, patients, and researchers across Nigerian that will support the prevention and management of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of generally good health or with hypertension

Exclusion Criteria:

* history of chronic diseases such as cardiovascular diseases (heart diseases), stroke, chronic kidney diseases, or pregnant or breastfeeding women, children below 18 years and adults above 70 years are also excluded from this study. Additionally, individuals who have made significant changes to their diet in the past six months or are currently following specific dietary restrictions will also be excluded from this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women deciding in Nigeria visiting River State University Teaching Hospital
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-07-23 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Validity of Clinical food frequency questionnaire (FFQ) | Phase 1 (4-8 weeks)
  Demonstrate the ability of a novel short clinical FFQ to accurately reflect diet habits
Feasibility of FFQ clinical tool in Nigerian clinic | Phase1 (4-8 weeks) and Phase 2 (4-8 weeks)
  Do patients, clinicians, and nurses see value in the tool in a clinical setting and accepting of it's use in the clinic

SECONDARY OUTCOMES:
Hypertension/Blood Pressure | Phase 2 (4 - 8 weeks)
  Association between FFQ clinical tool and blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zulyniak, PhD, Principal Investigator — University of Leeds
Locations (1):
- Royal State University, Port Harcourt, Nigeria

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data

REFERENCES:
- [Derived] Batubo NP, Auma CI, Moore JB, Zulyniak MA. Relative Validity and Reproducibility of a Dietary Screening Tool in Nigerian Health Care. Curr Dev Nutr. 2024 Sep 20;8(10):104459. doi: 10.1016/j.cdnut.2024.104459. eCollection 2024 Oct. PMID 39429509
- [Derived] Batubo NP, Nwanze NM, Alikor CA, Auma CI, Moore JB, Zulyniak MA. Empowering healthcare professionals in West Africa-A feasibility study and qualitative assessment of a dietary screening tool to identify adults at high risk of hypertension. PLoS One. 2024 Apr 25;19(4):e0294370. doi: 10.1371/journal.pone.0294370. eCollection 2024. PMID 38662712

DOCUMENTS (1):
  • Study Protocol (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/60/NCT05973760/Prot_000.pdf